CLINICAL TRIAL: NCT06713746
Title: Growth Differentiation Factor 15 Predictive Value, Prognostic Significance and Any Potential Correlation with Urea to Creatinine Ratio in Intensive Care Acquired Weakness
Brief Title: Growth Differentiation Factor 15 in ICU Acquired Muscle Weakness
Status: Completed | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Aya Hamdy Ahmed Nagy, Assistant lecturer of anesthesia and intensive care department, Minia University
Other Study IDs: 7292021
Record Dates: First submitted 2021-11-29; First posted 2024-12-03 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Muscle Weakness
Keywords: GDF15 Muscle weakness ICU
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ICU patients: muscle weakness
  Interventions: Diagnostic Test: growth differentiation factor 15

INTERVENTIONS:
Diagnostic Test: growth differentiation factor 15 — rowth differentiation factor-15 (GDF-15) is a novel cytokine secreted by a variety of cells like macrophages, adipocytes, normally expressed in high amounts by placenta
  Other Names: urea to creatinine ratio

SUMMARY:
Intensive care unit -acquired weakness (ICU- AW) is a common consequence linked to a worse outcome as evidenced by prolonged mechanical ventilation, longer ICU stays, greater mortality rates and a lower quality of life for survivors, so early detection and treatment of ICU-AW are critical. However, there is no "gold standard" currently available for assessing and diagnosing ICU-AW. It's crucial to develop diagnostic methods that enable for early detection and risk stratification in all critically ill patients, such as:

GDF-15 (growth differentiation factor-15) is thought to be a mediator of muscle atrophy because its level increases in the muscular atrophy As a result, measuring GDF-15 seems promise for diagnosing muscle atrophy.

DETAILED DESCRIPTION:
After obtaining the approval of research ethical committee of faculty of medicine, Minia university, written informed consent will be obtained from all participants or their legal representatives prior to study inclusion, this prospective cross sectional non randomized observational study will be conducted in intensive care unit Minia university hospital, on conscious non-mechanically ventilated patients with expected ICU stay 7 days or more during the period from January 2022 to December 2022. Based on inclusion and exclusion criteria, patients who met eligibility criteria, the prognosis and outcome of patients developing ICU-AW will be observed.

Parameters will be assessed:

1. Medical history, Age, gender, weight, BMI and APACHE II score ("Acute Physiology and Chronic Health Evaluation II") which is a severity-of-disease classification system one of several ICU scoring systems will be assessed in the day of admission.
2. SOFA score ("Sequential Organ Failure Assessment ") which will be assessed every day.
3. Routine lab investigations other than these in SOFA score as (Urea, Albumin, Hb, TLc, Pt, Ptt, RBG…..ect).
4. Urea:creatinine ratio: Urea and creatinine will be measured daily as a part of SOFA score and urea to creat will be calculated.
5. Plasma Growth differentiation 15 (GDF15) on 1, 4 and 7 days.
6. Ultrasound measurement of rectus femoris cross-sectional area (RFcsa) on 1, 4, 7, 10 and then every 3days according to patients stay in ICU.
7. Muscle Strength Assessment using the Medical Research Council (MRC) score on 1, 4 and 7 days where patients will be divided into an ICU-AW group and a non ICU-AW group according to their MRc-score on the 7th day.
8. Length of hospital and ICU stay.
9. Long term out come after 3 months survival, physical activity and return to work

ELIGIBILITY:
Inclusion Criteria:

* age more than 18 conscious patients patients with expected ICU stay more than 7 days

Exclusion Criteria:

- unconscious patients spinal cord injury limb fracture or amputations history of cognitive dysfunction severe oedema end stage kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients older than 18, conscious non mechanically ventilated patients and those with expected ICU stay more than 7 days during the period from September 2023 to September 2024
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Incidence | 1 year
  to investigate the incidence of intensive care unit acquired muscle weakness
Disease relations | 1 year
  to examine if there is any correlation between GDF15 level or urea-creatinine ratio and ICU acquired muscle weakness

SECONDARY OUTCOMES:
Daily activity and mortality | 1 year
  to investigate the influence of muscle weakness on daily activity and mortality of ICU acquired patients

CONTACTS AND LOCATIONS:
Locations (1):
- Minia university, Minya, Egypt